CLINICAL TRIAL: NCT06481839
Title: Impact of Starting Dose of Vasopressor on Hemodynamic Response in Shock
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Scott Benken, Clinical Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0748
Record Dates: First submitted 2024-06-24; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-dose NE (Active Comparator)
  Interventions: Other: Starting dose of NE
- High-dose NE (Active Comparator)
  Interventions: Other: Starting dose of NE

INTERVENTIONS:
Other: Starting dose of NE — Patients will be randomized to either low-dose (5mcg/min) or high-dose (15mcg/min) norepinephrine (NE) for their first vasopressor in shock.

SUMMARY:
This study is designed to assess the effect of initial vasopressor dose on clinical outcomes. To date, there are no clinical guidelines or recommendations regarding the dose of vasopressor medication that should be initiated before titrating to a mean arterial pressure (MAP) in patients with circulatory shock. High heterogeneity and clinical equipoise regarding this variable exist in routine clinical practice. However, there is strong evidence that delays in achieving MAP goals lead to worse clinical outcomes. The study will randomize patients with circulatory shock to a low (5mcg/min of norepinephrine) or high (15mcg/min of norepinephrine) initial starting dose followed by the usual protocolized titration to MAP goal. The time to reach the goal MAP, organ dysfunction, hospital length of stay, and mortality will be measured for each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old
* Patients who are diagnosed with shock (MAP < 65 mmHg) require the initiation of vasopressors
* Care provided in the ED or admission to the Medical Intensive Care Unit (MICU)
* Norepinephrine chosen as first-line vasopressor by the treating clinician

Exclusion Criteria:

* Patients who are receiving vasopressors or inotropes prior to UI Health hospital presentation/admission
* Baseline MAP >/= 65 mmHg
* Pregnant patients (checked as standard of care on admission)
* Prisoners.
* Immediate post-cardiac arrest patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-24 (Estimated); Primary Completion 2026-07-24 (Estimated); Study Completion 2028-07-24 (Estimated)

PRIMARY OUTCOMES:
Mean arterial blood pressure | During first shock episode, up to 28 days of shock episode.
  Time to achieve and sustain a mean arterial pressor greater than or equal to 65 mmHg

IPD SHARING:
Plan to Share IPD: No